CLINICAL TRIAL: NCT05019066
Title: The Effect of an Oral Herbal Combination Formulation on Hair Growth in Women With Self-perceived Hair Loss
Brief Title: Oral Herbal Combination Formulation and Hair Growth in Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided not to proceed with study.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1396273
Record Dates: First submitted 2021-08-04; First posted 2021-08-24 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Hair Loss; Hair Thinning
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal Combination Group (Active Comparator): * Tablets of the herbal formulation will be supplied from Banyan Botanicals (https://www.banyanbotanicals.com/healthy-hair-tablets-10)
  * Each 500 mg tablet contains a proprietary blend of: Eclipta alba, Emblica officinalis, Centella asiatica and Hibiscus sabdariffa
  * Dose: subjects in this group will take 2 herbal formulation tablets twice per day for a total of 4 tablets per day
  Interventions: Dietary Supplement: Herbal Supplementation
- Placebo Group (Placebo Comparator): * Supplement appearing similar to the herbal combination formulation.
  * Each placebo tablet will contain microcrystalline cellulose, dicalcium phosphate, PVPK30, sodium starch glycolate, magnesium stearate, OpaDry orange coating.
  * Dose: subjects in this group will take 2 placebo tablets twice per day for a total of 4 tablets per day
  Interventions: Dietary Supplement: Herbal Supplementation

INTERVENTIONS:
Dietary Supplement: Herbal Supplementation — A proprietary blend of: Eclipta alba, Emblica officinalis, Centella asiatica and Hibiscus sabdariffa.

SUMMARY:
The purpose of this research is to test the effects of an herbal combination formulation on hair growth in women with self-perceived hair loss.The information from this study may help to better understand how certain herbal supplements can affect hair growth. This may lead to better understanding of the hair, hair loss and help develop naturally-based treatment regimens in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Subject must be able to read and comprehend study procedures and consent forms.
* Women with self-perceived hair loss as confirmed by the investigator.
* Willing to maintain the same hairstyle, hair color, hair length and hair regimen throughout the study period. Subjects with color-treated hair will have the color treatment performed at the same time interval prior to each visit (if the color treatment was done 1 week prior to Visit 1, it should be repeated 1 week prior to Visit 2).
* Willing to keep diet and exercise routine consistent throughout study

Exclusion Criteria:

* Subjects should be generally healthy and have no smoking history in the past one year.
* Subjects must have no history of diabetes, metabolic syndrome, HIV, immune deficiency, autoimmune disease known cardiovascular disease, malignancy, kidney disease, or chronic steroid use.
* Women who are pregnant, planning to become pregnant or breastfeeding
* Those who are unable to discontinue medicated shampoos or topical scalp medications for two weeks prior to and during the study.
* Those who are unable to discontinue supplements containing Eclipta alba, Emblica officinalis, Centella asiatica and Hibiscus sabdariffa for one month prior to starting the study
* Those who have a known allergy to Eclipta alba, Emblica officinalis, Centella asiatica or Hibiscus sabdariffa
* Use of hair regrowth products in the previous 6 months
* Using or planned use of non-breathable wigs
* Those with a history of hair transplantation procedure
* Presence of other dermatological disorders causing alopecia
* Chemotherapy, radiation therapy or laser therapy (of scalp) in the last 6 months
* Light therapy in the past 3 months
* Participants using hormonal birth control unless on a stable / unchanged regimen for at least 3 months.
* Systemic treatment during the last 3 months before study inclusion that could interfere with the study medications (ie, minoxidil, corticosteroids, Aminexil, topical estrogens, ketoconazole, beta blocker, cimetidine, diazoxide, isotretinoin or vitamin A intake >10,000 IU/d)
* Use of ocular prostaglandins for less than 4 months before first study visit
* Those that are prisoners or cognitively impaired

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with self-perceived hair loss as confirmed by the investigator.
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-02-22 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Scalp photography Microscopic evaluation of hair Trichometry using the HairCheck© device | 24 weeks
  The HairCheck Trichometer will be used to measure hair caliber and hair density together and expresses them as a single number called the Hair Mass Index (HMI) or "Hair Number." The hair mass index (HMI) is ratio of the cross-sectional area of an isolated bundle of hair and the pre-measured area of skin from which it was taken using the trichometer device.
  The Folliscope (LeadM Corp, Seoul, South Korea)a phototrichogram device.5 will be used to measure density and hair diameter (per/cm2).

SECONDARY OUTCOMES:
Global Hair Growth and Global Hair Quality Assessment by investigator Hair Loss Subjective Questionnaire Symptom questionnaire | 24-weeks